CLINICAL TRIAL: NCT02432066
Title: Effects of GTS-21 on Smoking Behavior and Neurocognitive Functions
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not started and participants were not enrolled
Sponsor: University of Florida (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB201500393; Nixon2015 (Other: Nixon); R21DA038286 (NIH)
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation | interventions — 3-(2,4-dimethoxybenzylidene)anabaseine; anabaseine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GTS-21 (Active Comparator): Participants in the GTS-21 arm will receive 150 mg/BID GTS-21 over the course of 7 weeks. All participants will receive repeated neurobehavioral testing, laboratory assessment of cardiovascular and liver function, and provide weekly updates regarding smoking behavior, mood states, and side effects.
  Interventions: Drug: GTS-21
- Placebo (Placebo Comparator): Participants in the Placebo arm will receive placebo compound twice daily over the course of 7 weeks. All participants will receive repeated neurobehavioral testing, laboratory assessment of cardiovascular and liver function, and provide weekly updates regarding smoking behavior, mood states, and side effects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GTS-21 — GTS-21 is a partial alpha7 nicotinic agonist. GTS-21 will be compounded by the UF investigational pharmacy, and administered orally.
  Other Names: 3-(2,4-dimethoxybenzylidene) anabaseine (DMXB-A)
  Arms: GTS-21
Drug: Placebo — Oral placebo pills, compounded by the UF investigational pharmacy
  Other Names: Placebo Comparator
  Arms: Placebo

SUMMARY:
Attempts to quit cigarette smoking are often accompanied by negative mood and problems in attention and memory. These effects, in turn, may contribute to smoking relapse. This exploratory/developmental project examines the effects of a novel medication, GTS-21, on individuals interested in smoking cessation. It is hypothesized that GTS-21 will reduce negative affect, improve cognition and/or reduce smoking relapse in healthy adult men and women who are chronic cigarette smokers.

DETAILED DESCRIPTION:
The project is a clinical trial assessing the effects of GTS-21 (an α7 nicotinic receptor partial agonist) on smoking, mood, neurocognition, and neurophysiology, in a small sample of chronic smokers who are currently healthy and interested in smoking cessation. Using a double-blind, placebo controlled, parallel group design, 54 (27 women) community smokers who have demonstrated a readiness to quit will participate over a 7 week active trial. Subjects will be randomly assigned to active drug or placebo groups. Across the study period, participants will undergo repeated neurobehavioral testing, laboratory assessments of cardiovascular and liver function, and provide weekly updates regarding smoking behavior, mood state and side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 12 years of education
* Must report typical daily smoking of > 10 cigarettes/day over the previous year
* Must report a history of at least 3 years of regular smoking
* Must provide carbon monoxide measures of at least 6.5 ppm
* Must report a willingness to quit smoking

Exclusion Criteria:

* Participants engaged in behavioral and/or nicotine replacement therapies, or assisted quit efforts, within previous 6 months.
* Must not meet criteria for other substance dependence or major psychiatric disorders.
* Must be absent chronic medical conditions that might jeopardize health and safety, confound data interpretation or that contraindicate the administration of compounds acting at nAChR sites. This list includes disorders with direct effects on neurologic function (e.g., seizure disorders, transient ischemic events, chronic or active hepatic disease), metabolic disorders (e.g., uncontrolled Type 2 diabetes), or cardiovascular disease (e.g., hypertension, mitral valve compromise, tachycardia, or irregular heart rates).
* Must not smoke only cigars, pipes or hookahs or use nicotine products but not cigarettes
* Must not report current use of nicotine replacement therapies (i.e., occasions of > 4 h/week during a typical week, even if not used as a cessation aid)
* Must not have used bupropion within the previous year
* Must not report any past use (regardless of year) of varenicline
* Women may not be breastfeeding, pregnant or intending to become pregnant during the study period

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-29 (Estimated); Primary Completion 2018-12-29 (Estimated); Study Completion 2020-12-29 (Estimated)

PRIMARY OUTCOMES:
Change in Reported Nicotine Use from baseline at weeks 1, 2, 3, 4, 5, 6, 7, 8 | Change in baseline at Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  Nicotine use will be assessed using Timeline Followback procedures. Nicotine use will be reported to a trained interviewer using a Timeline Followback calendar, facilitated by calendars distributed to participants.
Change in Carbon Monoxide (CO) from baseline at weeks 5, 8 | Change in baseline at Week 5, Week 8
  Expired Carbon Monoxide levels will be quantified in parts per million.
Change in Urine Cotinine (COT) from baseline at weeks 5, 8 | Change in baseline at Week 5, Week 8
  Cotinine excreted in urine will be quantified in ng/mL

SECONDARY OUTCOMES:
Change in Beck Depression Inventory - II (BDI-II) from baseline at weeks 5, 8 | Change in baseline at Week 5, Week 8
  The Beck Depression Inventory will be used to quantify depressive symptomatology. The measure is a 21-item, self-report, multiple-choice inventory, with scores ranging from 0-63.
Change in State Anxiety Inventory (AI) from baseline at weeks 5, 8 | Change in baseline at Week 5, Week 8
  The State Anxiety Inventory will be used to quantify anxiety symptomatology. The measure is a 20-item, self-report, multiple-choice inventory, with scores ranging from 20-80.
Change in State Anger (ANG-S) from baseline at weeks 5, 8 | Change in baseline at Week 5, Week 8
  The Spielberger State Anger Inventory will be used to assess state anger. The measure is a 20-item, self-report, multiple-choice inventory, with scores ranging from 20-80.
Pill Count - Week 1 | Week 1
  Medication compliance will be assessed with pill counts.
Pill Count - Week 5 | Week 5
  Medication compliance will be assessed with pill counts.
Pill Count - Week 8 | Week 8
  Medication compliance will be assessed with pill counts.
Change in Minnesota Withdrawal Scale from baseline at weeks 1, 2, 3, 4, 5, 6, 7, 8 | Change in baseline at Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  The Minnesota Withdrawal Scale measures self-reported severity of nicotine withdrawal. The measure has 15 items, with five possible responses (0-5), thus scores on the scale range from 0 to 60.
Systematic Assessment for Treatment Emergent Events (SAFTEE) - Week 1 | Week 1
  The SAFTEE assesses potential side effects across a broad range of potential somatic effects. The measure includes 132 potential areas in which participants might report effects, including opportunities for the participant to describe otherwise unlisted option. Each area is scored on a 5-point scale.
Systematic Assessment for Treatment Emergent Events (SAFTEE) - Week 2 | Week 2
  The SAFTEE assesses potential side effects across a broad range of potential somatic effects. The measure includes 132 potential areas in which participants might report effects, including opportunities for the participant to describe otherwise unlisted option. Each area is scored on a 5-point scale.
Systematic Assessment for Treatment Emergent Events (SAFTEE) - Week 3 | Week 3
  The SAFTEE assesses potential side effects across a broad range of potential somatic effects. The measure includes 132 potential areas in which participants might report effects, including opportunities for the participant to describe otherwise unlisted option. Each area is scored on a 5-point scale.
Systematic Assessment for Treatment Emergent Events (SAFTEE) - Week 4 | Week 4
  The SAFTEE assesses potential side effects across a broad range of potential somatic effects. The measure includes 132 potential areas in which participants might report effects, including opportunities for the participant to describe otherwise unlisted option. Each area is scored on a 5-point scale.
Systematic Assessment for Treatment Emergent Events (SAFTEE) - Week 5 | Week 5
  The SAFTEE assesses potential side effects across a broad range of potential somatic effects. The measure includes 132 potential areas in which participants might report effects, including opportunities for the participant to describe otherwise unlisted option. Each area is scored on a 5-point scale.
Systematic Assessment for Treatment Emergent Events (SAFTEE) - Week 6 | Week 6
  The SAFTEE assesses potential side effects across a broad range of potential somatic effects. The measure includes 132 potential areas in which participants might report effects, including opportunities for the participant to describe otherwise unlisted option. Each area is scored on a 5-point scale.
Systematic Assessment for Treatment Emergent Events (SAFTEE) - Week 7 | Week 7
  The SAFTEE assesses potential side effects across a broad range of potential somatic effects. The measure includes 132 potential areas in which participants might report effects, including opportunities for the participant to describe otherwise unlisted option. Each area is scored on a 5-point scale.
Systematic Assessment for Treatment Emergent Events (SAFTEE) - Week 8 | Week 8
  The SAFTEE assesses potential side effects across a broad range of potential somatic effects. The measure includes 132 potential areas in which participants might report effects, including opportunities for the participant to describe otherwise unlisted option. Each area is scored on a 5-point scale.
Change in Profile of Mood States 2-A from Baseline at Week 1, 2, 3, 4, 5, 6, 7, 8 | Change in baseline at Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  The Profile of Mood States-2 (short-form for adults) The POMS 2 is a multi-dimensional, assessment of transient moods, and states of affect. The measure includes 35 items, each rated on a 5-point scale (0-4).
Rapid Visual Information Processing task (Behavior) - Baseline | Baseline
  The Rapid Visual Information Processing task is an attention task. Subjects are instructed to detect and respond as quickly, yet as accurately, as possible when a target of three consecutive odd or even digits are presented. Digits are presented at the rate of approximately 100 per minute. Hits are separated by a varying number of stimuli (e.g., between 5 and 30 digits). Dependent variables will include accuracy and reaction time.
Rapid Visual Information Processing task - (Behavior) - Week 8 | Week 8
  The Rapid Visual Information Processing task is an attention task. Subjects are instructed to detect and respond as quickly, yet as accurately, as possible when a target of three consecutive odd or even digits are presented. Digits are presented at the rate of approximately 100 per minute. Hits are separated by a varying number of stimuli (e.g., between 5 and 30 digits). Dependent variables will include accuracy and reaction time.
Rapid Visual Information Processing task - (EEG) - Baseline | Baseline
  The Rapid Visual Information Processing task is an attention task. Subjects are instructed to detect and respond as quickly, yet as accurately, as possible when a target of three consecutive odd or even digits are presented. Digits are presented at the rate of approximately 100 per minute. Hits are separated by a varying number of stimuli (e.g., between 5 and 30 digits). Dependent variables will include electrophysiological measures gathered during task participation, including the peak and latency of the P3, P2, and N1 components.
Rapid Visual Information Processing task - (EEG) - Week 8 | Week 8
  The Rapid Visual Information Processing task is an attention task. Subjects are instructed to detect and respond as quickly, yet as accurately, as possible when a target of three consecutive odd or even digits are presented. Digits are presented at the rate of approximately 100 per minute. Hits are separated by a varying number of stimuli (e.g., between 5 and 30 digits). Dependent variables will include electrophysiological measures gathered during task participation, including the peak and latency of the P3, P2, and N1 components.
Measurement of GTS-21 Concentration in Blood - Week 5 | Week 5
  Blood samples will be collected and analyzed for their concentration of GTS-21.
Measurement of GTS-21 Concentration in Blood - Week 8 | Week 8
  Blood samples will be collected and analyzed for their concentration of GTS-21.
Trail Making Test A (TMT-A) - Baseline | Baseline
  The Trail Making Test A consists of numbered 25 circles distributed over a sheet of paper. Participants draw a line between consecutive circles as quickly and accurately as possible. The dependent variable is time to completion of the task.
Trail Making Test A (TMT-A) - Week 5 | Week 5
  The Trail Making Test A consists of numbered 25 circles distributed over a sheet of paper. Participants draw a line between consecutive circles as quickly and accurately as possible. The dependent variable is time to completion of the task.
Trail Making Test A (TMT-A) - Week 8 | Week 8
  The Trail Making Test A consists of numbered 25 circles distributed over a sheet of paper. Participants draw a line between consecutive circles as quickly and accurately as possible. The dependent variable is time to completion of the task.
Trail Making Test B (TMT-B) - Baseline | Baseline
  The Trail Making Test B consists of 25 circles distributed over a sheet of paper, labeled with numbers (1-13) and letters (A-L). Participants draw a line between circles, alternating between consecutive numbers and letters (i.e., 1 to A, A to 2, 2 to B, etc.) as quickly and accurately as possible. The dependent variable is time to completion of the task.
Trail Making Test B (TMT-B) - Week 5 | Week 5
  The Trail Making Test B consists of 25 circles distributed over a sheet of paper, labeled with numbers (1-13) and letters (A-L). Participants draw a line between circles, alternating between consecutive numbers and letters (i.e., 1 to A, A to 2, 2 to B, etc.) as quickly and accurately as possible. The dependent variable is time to completion of the task.
Trail Making Test B (TMT-B) - Week 8 | Week 8
  The Trail Making Test B consists of 25 circles distributed over a sheet of paper, labeled with numbers (1-13) and letters (A-L). Participants draw a line between circles, alternating between consecutive numbers and letters (i.e., 1 to A, A to 2, 2 to B, etc.) as quickly and accurately as possible. The dependent variable is time to completion of the task.
N-Back Working Memory Task (Behavior) - Baseline | Baseline
  The 'n-back' test is a measure of working memory entailing the presentation of a stream of numbers, presented singly, and separated by neutral stimuli (i.e., "+"). Ss press a button when the presented stimulus is the same as the one that occurred 'n-back', i.e., some specific number back. The 'n-back' will vary across blocks (i.e., 1 or 2 back). A control condition, requiring Ss to press the button when a blank slide appears, will also be employed. Dependent variables will include accuracy and reaction time.
N-Back Working Memory Task (Behavior) - Week 8 | Week 8
  The 'n-back' test is a measure of working memory entailing the presentation of a stream of numbers, presented singly, and separated by neutral stimuli (i.e., "+"). Ss press a button when the presented stimulus is the same as the one that occurred 'n-back', i.e., some specific number back. The 'n-back' will vary across blocks (i.e., 1 or 2 back). A control condition, requiring Ss to press the button when a blank slide appears, will also be employed. Dependent variables will include accuracy and reaction time.
N-Back Working Memory Task (EEG) - Baseline | Baseline
  The 'n-back' test is a measure of working memory entailing the presentation of a stream of numbers, presented singly, and separated by neutral stimuli (i.e., "+"). Ss press a button when the presented stimulus is the same as the one that occurred 'n-back', i.e., some specific number back. The 'n-back' will vary across blocks (i.e., 1 or 2 back). A control condition, requiring Ss to press the button when a blank slide appears, will also be employed. Dependent variables will include electrophysiological measures gathered during task participation, including the peak and latency of the P3, P2, and N1 components.
N-Back Working Memory Task (EEG) - Week 8 | Week 8
  The 'n-back' test is a measure of working memory entailing the presentation of a stream of numbers, presented singly, and separated by neutral stimuli (i.e., "+"). Ss press a button when the presented stimulus is the same as the one that occurred 'n-back', i.e., some specific number back. The 'n-back' will vary across blocks (i.e., 1 or 2 back). A control condition, requiring Ss to press the button when a blank slide appears, will also be employed. Dependent variables will include electrophysiological measures gathered during task participation, including the peak and latency of the P3, P2, and N1 components.
Simple Reaction Time Test - Baseline | Baseline
  In this computerized task, subjects must press a button as quickly as possible each time a designed symbol appears on the screen. This test serves as a perceptual-motor control. The dependent measure is reaction time.
Simple Reaction Time Test - Week 5 | Week 5
  In this computerized task, subjects must press a button as quickly as possible each time a designed symbol appears on the screen. This test serves as a perceptual-motor control. The dependent measure is reaction time.
Simple Reaction Time Test - Week 8 | Week 8
  In this computerized task, subjects must press a button as quickly as possible each time a designed symbol appears on the screen. This test serves as a perceptual-motor control. The dependent measure is reaction time.
Little Man Test - Baseline | Baseline
  In this computerized mental rotation test, subjects must indicate the hand in which a simulated figure holds an object. The dependent measures are accuracy and reaction time.
Little Man Test - Week 8 | Week 8
  In this computerized mental rotation test, subjects must indicate the hand in which a simulated figure holds an object. The dependent measures are accuracy and reaction time.
Visual-Perceptual Analysis Test - Baseline | Baseline
  In this computerized task, subjects must distinguish which of three similar shapes differs from the other two. Dependent measures include accuracy and reaction time.
Visual-Perceptual Analysis Test - Week 5 | Week 5
  In this computerized task, subjects must distinguish which of three similar shapes differs from the other two. Dependent measures include accuracy and reaction time.
Visual-Perceptual Analysis Test - Week 8 | Week 8
  In this computerized task, subjects must distinguish which of three similar shapes differs from the other two. Dependent measures include accuracy and reaction time.
Wisconsin Card Sorting Test - Baseline | Baseline
  The Wisconsin Card Sort Test is a computerized task which requires subjects to match "cards" based on shifting matching rules which include color, shape, and number of symbols. The dependent measures for this task include accuracy and response time.
Wisconsin Card Sorting Test - Week 8 | Week 8
  The Wisconsin Card Sort Test is a computerized task which requires subjects to match "cards" based on shifting matching rules which include color, shape, and number of symbols. The dependent measures for this task include accuracy and response time.
Sternberg Short-Term Memory Test - Baseline | Baseline
  The Sternberg Short-Term Memory Test is a computerized task in which participants are shown four digits, presented one at a time, followed by a probe digit. They must determine if the probe digit was in the original set of digits, and recall the digits. The dependent variables are probe accuracy, number of correct recalls, and time to completion.
Sternberg Short-Term Memory Test - Week 8 | Week 8
  The Sternberg Short-Term Memory Test is a computerized task in which participants are shown four digits, presented one at a time, followed by a probe digit. They must determine if the probe digit was in the original set of digits, and recall the digits. The dependent variables are probe accuracy, number of correct recalls, and time to completion.
Stroop Color Word Task - Baseline | Baseline
  The Stroop Task is a measure of inhibitory control. Subjects are directed to name the colors words are printed in (i.e., "blue"), while ignoring the incongruent meaning of the words. The dependent measures include number correct and number completed.
Stroop Color Word Task - Week 8 | Week 8
  The Stroop Task is a measure of inhibitory control. Subjects are directed to name the colors words are printed in (i.e., "blue"), while ignoring the incongruent meaning of the words. The dependent measures include number correct and number completed.
Digit Symbol Substitution Task - Baseline | Baseline
  The Digit Symbol Substitution Task requires attention and set-switching. Subjects must translate between numbers and symbols, using a key provided. The dependent measure is number of correct responses completed.
Digit Symbol Substitution Task - Week 5 | Week 5
  The Digit Symbol Substitution Task requires attention and set-switching. Subjects must translate between numbers and symbols, using a key provided. The dependent measure is number of correct responses completed.
Digit Symbol Substitution Task - Week 8 | Week 8
  The Digit Symbol Substitution Task requires attention and set-switching. Subjects must translate between numbers and symbols, using a key provided. The dependent measure is number of correct responses completed.
Metabolic Panel - Baseline | Baseline
  Liver Function Test will measure a standard array of blood chemistries, including electrolytes, blood glucose, protein, liver enzymes (aminotransferase/alanine aminotransferase), bilirubin, creatinine, and blood urea nitrogen.
Metabolic Panel - Week 2 | Week 2
  Liver Function Test will measure a standard array of blood chemistries, including electrolytes, blood glucose, protein, liver enzymes (aminotransferase/alanine aminotransferase), bilirubin, creatinine, and blood urea nitrogen.
Metabolic Panel - Week 5 | Week 5
  Liver Function Test will measure a standard array of blood chemistries, including electrolytes, blood glucose, protein, liver enzymes (aminotransferase/alanine aminotransferase), bilirubin, creatinine, and blood urea nitrogen.
Metabolic Panel - Week 8 | Week 8
  Liver Function Test will measure a standard array of blood chemistries, including electrolytes, blood glucose, protein, liver enzymes (aminotransferase/alanine aminotransferase), bilirubin, creatinine, and blood urea nitrogen.
Metabolic Panel - Week 9 (Followup) | Week 9
  Liver Function Test will measure a standard array of blood chemistries, including electrolytes, blood glucose, protein, liver enzymes (aminotransferase/alanine aminotransferase), bilirubin, creatinine, and blood urea nitrogen.
Urinalysis - Baseline | Baseline
  Standard urinalysis will be conducted, including urine pH, red cell count, white cell count, specific gravity, and bacteria content.
Urinalysis - Week 2 | Week 2
  Standard urinalysis will be conducted, including urine pH, red cell count, white cell count, specific gravity, and bacteria content.
Urinalysis - Week 5 | Week 5
  Standard urinalysis will be conducted, including urine pH, red cell count, white cell count, specific gravity, and bacteria content.
Urinalysis - Week 8 | Week 8
  Standard urinalysis will be conducted, including urine pH, red cell count, white cell count, specific gravity, and bacteria content.
Urinalysis - Week 9 (Followup) | Week 9
  Standard urinalysis will be conducted, including urine pH, red cell count, white cell count, specific gravity, and bacteria content.
Electrocardiogram - Baseline | Baseline
  Standard electrocardiographic data will be collected, including heart rate (BPM) and time between start of the Q wave and end of the T wave (QT interval).
Electrocardiogram - Week 1 | Week 1
  Standard electrocardiographic data will be collected, including heart rate (BPM) and time between start of the Q wave and end of the T wave (QT interval).
Change in Reported Drug and Alcohol Use from baseline at weeks 1, 2, 3, 4, 5, 6, 7, 8 | Change in baseline at Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8
  Drug and alcohol use will be assessed using Timeline Followback procedures. Drug and alcohol use will be reported to a trained interviewer using a Timeline Followback calendar, facilitated by calendars distributed to participants.
Change in Blood Pressure from baseline at weeks 2, 5, 8, 9 | Change in baseline at Week 2, Week 5, Week 8, Week 9
  Systolic and Diastolic pressures will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Nixon, PhD, Principal Investigator — University of Florida